CLINICAL TRIAL: NCT02545621
Title: A Role for RAGE/TXNIP/Inflammasome Axis in Alveolar Macrophage Activation During ARDS (RIAMA): a Proof-of-concept Clinical Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0243
Record Dates: First submitted 2015-09-08; First posted 2015-09-10 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2016-07

CONDITIONS: Acute Respiratory Distress Syndrome; Mechanical Ventilation
Keywords: Receptor for advanced glycation end products (RAGE); Acute respiratory distress syndrome (ARDS); Monocyte/Macrophage activation; Fluorescence-Activated Cell Sorting (FACS) analysis; Thioredoxin interacting protein (TXNIP); NOD-like receptor family, pyrin domain containing 3 (NLRP3); Inflammasome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- ARDS Group (acute respiratory distress syndrome): The purpose of this monocentric observational prospective pathophysiology study is to compare alveolar monocyte/macrophage activation profiles between patients with or without ARDS
  Interventions: Other: RAGE TXNIP Inflammasome axis
- control group: The purpose of this monocentric observational prospective pathophysiology study is to compare alveolar monocyte/macrophage activation profiles between patients with or without ARDS
  Interventions: Other: RAGE TXNIP Inflammasome axis

INTERVENTIONS:
Other: RAGE TXNIP Inflammasome axis

SUMMARY:
RAGE (the receptor for advanced glycation end-products) is a marker of alveolar type I cell injury and a pivotal mediator of acute inflammation and innate immunity. RAGE pathway is highly regulated; the interaction of the transmembrane receptor with its various ligands (e.g. HMGB1, S100A12) ultimately leads to NF-kB activation and RAGE upregulation itself, but precise RAGE functions and intracellular pathways remain underexplored. During ARDS, monocyte and macrophage activation could modulate alveolar inflammation and repair.

As RAGE is also expressed at the surface of monocytes/macrophages, we hypothesize that alveolar monocyte/macrophage activation may be mediated through a RAGE-TXNIP (thioredoxin interacting protein)-NLRP3/inflammasome intracellular pathway. The purpose of this observational prospective study is to compare alveolar monocyte/macrophage activation profiles (as assessed by Fluorescence-Activated Cell Sorting (FACS)) in mechanically ventilated patients with or without ARDS.

DETAILED DESCRIPTION:
BACKGROUND:

The receptor for advanced glycation end products (RAGE) was recently identified as a promising new marker of alveolar type I cell injury. RAGE is a member of the immunoglobulin superfamily that acts as a multiligand receptor and is involved in propagating inflammatory responses in various cell populations. While the precise function of RAGE remains unclear, the elevated levels of RAGE, and its soluble isoform sRAGE, correlate with severity of acute respiratory distress syndrome (ARDS) in human and animal studies.

RAGE pathway is highly regulated; the interaction of the transmembrane receptor with its various ligands (e.g. HMGB1, S100A12) ultimately leads to NF-kB activation and RAGE upregulation itself. During ARDS, monocyte and macrophage activation could modulate alveolar inflammation and repair. As RAGE is also expressed at the surface of monocytes/macrophages, we hypothesize that alveolar monocyte/macrophage activation may be mediated through a RAGE-TXNIP (thioredoxin interacting protein)-NLRP3/inflammasome intracellular pathway.

DESIGN NARRATIVE:

The purpose of this monocentric observational prospective pathophysiology study is to compare alveolar monocyte/macrophage activation profiles between patients with or without ARDS.

Using Fluorescence-Activated Cell Sorting (FACS) analysis, monocyte/macrophage activation profiles will be characterized in patients within the first 24 hours after onset of ARDS and in matched mechanically ventilated controls. Markers of M1 ("pro-inflammatory") or M2 ("anti-inflammatory") activation, along with RAGE, TXNIP, NLRP3 FACS labeling in alveolar monocytes/macrophages will be analyzed along with protein measurements (IL-1β, TXNIP, NLRP3, sRAGE, HMGB1, S100A12) in the bronchoalveolar lavage fluid.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients without ARDS and under mechanical ventilation for less than 24 hours
* Patients within the first 24 hours after onset of moderate to severe ARDS according to the 2012 Berlin definition (ARDS group)

Exclusion Criteria:

* - Pregnancy
* Acute exacerbation of diabetes (ketoacidosis, hyperosmolar hyperglycemic state)
* Patient under mechanical ventilation for > 7 days
* Dialysis-dependent chronic renal failure
* Alzheimer's disease
* Amyloidosis
* Evolutive neoplastic lesion
* Chronic pulmonary disease requiring long-term oxygen therapy or mechanical ventilation
* Chemotherapy treatment in the last 30 days
* Severe neutropenia (<0.5 G/l)

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients without ARDS and under mechanical ventilation for less than 24 hours
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
FACS analysis of RAGE-TXNIP-NLRP3 pathway in alveolar monocytes/macrophages | at day1
  FACS analysis of RAGE-TXNIP-NLRP3 pathway in alveolar monocytes/macrophages from patients within the first 24 hours after onset of ARDS (ARDS group) and from sex- and age-matched mechanically ventilated controls (control group)

SECONDARY OUTCOMES:
- FACS analysis of M1 ("pro-inflammatory") and M2 ("anti-inflammatory") markers | at baseline
  - FACS analysis of M1 ("pro-inflammatory") and M2 ("anti-inflammatory") markers (e.g., CD45, CD16, CD14, CD163, CD206, ICAM-1) in alveolar monocytes/macrophages from patients from both groups at baseline
IL-1β, TXNIP, NLRP3, sRAGE, HMGB1, S100A12 measurements | at baseline
  - IL-1β, TXNIP, NLRP3, sRAGE, HMGB1, S100A12 measurements (duplicate ELISA) in the bronchoalveolar lavage fluid from patients from both groups at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu JABAUDON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France